CLINICAL TRIAL: NCT02431923
Title: Partnership for Research on Ebola Virus (PREVAIL) Prevail III: Ebola Natural History Study
Brief Title: Ebola Virus Disease Survivors: Clinical and Immunologic Follow-up
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 150122; 15-I-0122
Record Dates: First submitted 2015-04-30; First posted 2015-05-01 (Estimated); Last update posted 2022-10-10 (Actual); Status verified 2022-10

CONDITIONS: Ebola Virus Disease
Keywords: Sequelae; Seroprevalence; Household Contacts; Natural History
MeSH Terms: conditions — Hemorrhagic Fever, Ebola

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- EVD Close Contacts: At least one of the following:-Household contact of survivor at time of or since EVD event-Sexual contact with survivor since EVD event-Other selected contacts
- EVD Survivors: Subject listed on the Ministry of Health registry for Ebola survivors
- Non Contact Controls: Selected Controls

SUMMARY:
Background:

- Ebola is a lethal disease. A lot is still unknown about Ebola and its long-term effects. Researchers want to learn what ill health conditions Ebola survivors have. They want to learn if Ebola survivors can infect others in their household through close contact. They also want to learn if Ebola survivors are immune from getting Ebola again. To learn these things, they want to follow people in Liberia for 5 years.

Objectives:

- To learn how Ebola affects the health of survivors and the people they live with.

Eligibility:

- People in Liberia who had Ebola in the past 2 years, who share a household with someone who had Ebola, or who got ill and went to an Ebola Treatment Unit but were sent home because they did not have Ebola.

Design:

* Participants will be screened with family illness history, physical exam, and blood tests. They may have an eye exam.
* Ebola survivors and those who went to a Treatment Unit but did not have Ebola will visit a clinic at 3, 6, and 12 months, then every 6 months for 5 years. At each visit, they will repeat the screening tests.
* Participants who live with someone who had Ebola will have only the screening visit. But they may be asked to return for follow-up visits. These visits will help researchers learn more about the differences between those who have had Ebola and those who have not.
* Participants brought to the NIH Clinical Center will have documentation of positive Ebola virus PCR and a clinical syndrome compatible with acute EVD.
* The study will last 5 years.

DETAILED DESCRIPTION:
Between 1994 and the present, there have been several Ebola virus outbreaks affecting mostly countries in Central Africa. However, the 2014 West African outbreak significantly exceeds all previous outbreaks in geographic range and number of individuals affected. Ebola virus disease (EVD) is highly lethal with case fatality rates of 70-80% in the current West African outbreak. While the clinical manifestations of acute Ebola virus infection are well documented, little is known about long-term sequelae, ability to transmit Ebola, or long-term protective immunity in survivors from EVD. The purpose of this protocol is to study these questions in a cohort of EVD survivors from Liberia.

ELIGIBILITY:
* INCLUSION CRITERIA FOR EVD SURVIVORS

A volunteer of any age with a diagnosis of EVD within the past 2 years who is on the Ministry of Health (MOH) Registry of EVD survivors is eligible to participate.

* Willingness to participate in examinations at one of the participating health facilities
* Willingness to provide informed consent/assent

Individuals on the MOH Registry were PCR positive for EVD and treated at an Ebola Treatment Unit (ETU), Community Care Center (CCC) or holding center. Periodically, participants enrolled will be matched against the MOH Registry to verify that those enrolled are EVD survivors. If a participant enrolled is not on the registry, their antibody levels at baseline will be assessed. If antibody levels are present, the participant will continue to be followed as an EVD survivor. If antibody levels are not present, the participants will no longer be followed as an EVD survivor and may be withdrawn from the study. Participants brought to the NIH Clinical Center will have documentation of positive Ebola virus PCR and a clinical syndrome compatible with acute EVD.

EXCLUSION CRITERION FOR EVD SURVIVORS

Any condition in the judgment of the study staff that would make the volunteer unable to participate in the study.

Max Age: 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Survivors of EVD, household contacts, non EVD Controls
Sampling Method: Non-Probability Sample
Enrollment: 4043 (Actual)
Dates: Start 2017-12-02 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
To characterize the clinical sequelae seen in convalescent Ebola virus disease (EVD) patients. | Throughout
  longterm sequelae, ability to transmit Ebola, or long-term protective immunity in survivors convalescing from EVD
Assess whether convalescent EVD patients can transmit infection to household and sexual contacts as determined by development of EVD or Ebola seroconversion in contacts | Throughout
  longterm sequelae, ability to transmit Ebola, or long-term protective immunity in survivors convalescing from EVD

SECONDARY OUTCOMES:
Better define the immune response in EVD survivors. | Throughout
  longterm sequelae, ability to transmit Ebola, or long-term protective immunity in survivors convalescing from EVD

CONTACTS AND LOCATIONS:
Overall Officials: Michael C Sneller, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (4):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States
- Liberia (3):
  - CH Rennie Hospital, Kakata
  - Duport Clinic, Monrovia
  - JFK Hospital, Monrovia

REFERENCES:
- [Background] Rowe AK, Bertolli J, Khan AS, Mukunu R, Muyembe-Tamfum JJ, Bressler D, Williams AJ, Peters CJ, Rodriguez L, Feldmann H, Nichol ST, Rollin PE, Ksiazek TG. Clinical, virologic, and immunologic follow-up of convalescent Ebola hemorrhagic fever patients and their household contacts, Kikwit, Democratic Republic of the Congo. Commission de Lutte contre les Epidemies a Kikwit. J Infect Dis. 1999 Feb;179 Suppl 1:S28-35. doi: 10.1086/514318. PMID 9988162
- [Background] Kibadi K, Mupapa K, Kuvula K, Massamba M, Ndaberey D, Muyembe-Tamfum JJ, Bwaka MA, De Roo A, Colebunders R. Late ophthalmologic manifestations in survivors of the 1995 Ebola virus epidemic in Kikwit, Democratic Republic of the Congo. J Infect Dis. 1999 Feb;179 Suppl 1:S13-4. doi: 10.1086/514288. PMID 9988158
- [Derived] Postnikova EN, Pettitt J, Van Ryn CJ, Holbrook MR, Bollinger L, Yu S, Cai Y, Liang J, Sneller MC, Jahrling PB, Hensley LE, Kuhn JH, Fallah MP, Bennett RS, Reilly C. Scalable, semi-automated fluorescence reduction neutralization assay for qualitative assessment of Ebola virus-neutralizing antibodies in human clinical samples. PLoS One. 2019 Aug 27;14(8):e0221407. doi: 10.1371/journal.pone.0221407. eCollection 2019. PMID 31454374
- [Derived] PREVAIL III Study Group; Sneller MC, Reilly C, Badio M, Bishop RJ, Eghrari AO, Moses SJ, Johnson KL, Gayedyu-Dennis D, Hensley LE, Higgs ES, Nath A, Tuznik K, Varughese J, Jensen KS, Dighero-Kemp B, Neaton JD, Lane HC, Fallah MP. A Longitudinal Study of Ebola Sequelae in Liberia. N Engl J Med. 2019 Mar 7;380(10):924-934. doi: 10.1056/NEJMoa1805435. PMID 30855742
- [Derived] Kelly JD, Weiser SD, Wilson B, Cooper JB, Glayweon M, Sneller MC, Drew C, Steward WT, Reilly C, Johnson K, Fallah MP. Ebola virus disease-related stigma among survivors declined in Liberia over an 18-month, post-outbreak period: An observational cohort study. PLoS Negl Trop Dis. 2019 Feb 27;13(2):e0007185. doi: 10.1371/journal.pntd.0007185. eCollection 2019 Feb. PMID 30811388
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2015-I-0122.html